CLINICAL TRIAL: NCT06070675
Title: Comparison of a Paper and Automated Bladder Diary in Pediatric Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Lola Bladt, Sub-Investigator, Universiteit Antwerpen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: BUN B3002023000056
Record Dates: First submitted 2023-09-18; First posted 2023-10-06 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Lower Urinary Tract Symptoms; Voiding Disorders; Enuresis; Overactive Bladder
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Enuresis; Urinary Bladder, Overactive

STUDY DESIGN:
Intervention Model Description: Mixed methods, randomized 2x2 crossover trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paper bladder diary (pBD) (Other): Patients will complete the paper bladder diary at home for at least 2 consecutive days.
  Interventions: Other: Paper bladder diary
- Automated bladder diary (autoBD) (Other): Patients will complete the automated bladder diary (Minze Diary Pod) at home for at least 2 consecutive days.
  Interventions: Device: Minze Diary Pod

INTERVENTIONS:
Device: Minze Diary Pod — The automated bladder diary utilized in this study consists of the Minze Diary Pod and Minze Flow app. The Diary Pod is a capacitance-based measuring device, that automatically registers voided volumes and time of void. The Diary Pod connects via Bluetooth to the Minze Flow app to request additional information from the patient, such as urge, drinks and leakages.
  Arms: Automated bladder diary (autoBD)
Other: Paper bladder diary — The paper bladder diary utilized in this study is a paper timetable that has the patient enter (in the columns of the timetable) drinks in ml, urinations in ml (using a measuring cup) and leakage episodes for the nearest hours (rows of the timetable).
  Arms: Paper bladder diary (pBD)

SUMMARY:
The purpose of this study is to compare an automated bladder diary (autoBD) to a paper bladder diary (pBD) on their level of agreement, patient compliance and satisfaction. It is a mixed methods, randomized 2x2 crossover trial. Pediatric patients (6 to 12 years) presenting to the clinic and identified as requiring a bladder diary will be recruited. Participants will be randomized either to group 1, where they complete the paper bladder diary (pBD) and then the automated bladder diary (autoBD), or to group 2, where they complete the autoBD and then the pBD. Both diaries are kept for at least 2 consecutive days with a wash-out period of 2 to 6 days between the two diaries. Mean differences and the level of agreement between the pBD and autoBD will be analysed using Bland Altman plots for key diary parameters.

After completion of each diary format, participants will complete a short online survey regarding compliance, satisfaction and their preference, if any. Finally, a selection of participants and their parents will be invited for an open-ended interview.

The participating healthcare professionals will be asked to score each pBD and autoBD on patient compliance when processing the diary. Furthermore, surveys and open-ended interviews will be conducted to assess their overall satisfaction of each diary type and their preference, if any.

DETAILED DESCRIPTION:
For some time now, patient compliance with paper bladder diaries is being questioned. Paper bladder diaries are often incomplete, unreliable and/or of low quality. Multiple electronic bladder diaries have been developed to overcome some of the limitations associated with paper bladder diaries. However, based on several comparison studies between paper and electronic bladder diaries, it is not clear whether an electronic format alone is truly superior to the paper format. The investigators want to introduce and evaluate the feasibility of a new type of bladder diary: an automated bladder diary. In contrast to an electronic diary, an automated diary automatically registers voiding data using a connected measuring device. An electronic diary simply eliminates the use of paper, but the patient still needs to measure the voided volumes with a urinary container and manually enter them in the electronic diary. The investigators believe an automated diary may lead to improved patient compliance by reducing the required efforts from the patient and instead provide guidance and prompts.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients presenting to the clinic and identified as requiring a bladder diary
* Age: 6 to 12 years
* Sex: male or female
* Child and/or parent own and are able to operate a smartphone and/or tablet

Exclusion Criteria:

* Change in urologic treatment during the data collection period
* Inability to hold the Diary Pod while urinating
* Inability to speak, read and write Dutch

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Level of agreement average daytime volume (ml) | Through study completion, an average of 1.5 year
  What are the mean differences and the limits of agreement between the pBD and autoBD for average daytime volume (ml).

SECONDARY OUTCOMES:
Level of agreement maximum voided volume (ml) | Through study completion, an average of 1.5 year
  What are the mean differences and the limits of agreement between the pBD and autoBD for maximum voided volume (ml).
Level of agreement 24h voided volume (ml) | Through study completion, an average of 1.5 year
  What are the mean differences and the limits of agreement between the pBD and autoBD for 24h voided volume (ml).
Level of agreement nighttime voided volume (ml) | Through study completion, an average of 1.5 year
  What are the mean differences and the limits of agreement between the pBD and autoBD for nighttime voided volume (ml).
Level of agreement average daytime volume versus age expected bladder capacity (%) | Through study completion, an average of 1.5 year
  What are the mean differences and the limits of agreement between the pBD and autoBD for average daytime volume versus age expected bladder capacity (%).
Level of agreement maximum voided volume versus age expected bladder capacity (%) | Through study completion, an average of 1.5 year
  What are the mean differences and the limits of agreement between the pBD and autoBD for maximum voided volume versus age expected bladder capacity (%).
Level of agreement nighttime voided volume versus age expected bladder capacity (%) | Through study completion, an average of 1.5 year
  What are the mean differences and the limits of agreement between the pBD and autoBD for nighttime voided volume versus age expected bladder capacity (%).
Level of agreement nighttime voided volume versus 24h voided volume (%) | Through study completion, an average of 1.5 year
  What are the mean differences and the limits of agreement between the pBD and autoBD for nighttime voided volume versus 24h voided volume (%).
Level of agreement nighttime voided volume versus daytime voiding frequency | Through study completion, an average of 1.5 year
  What are the mean differences and the limits of agreement between the pBD and autoBD for nighttime voided volume versus daytime voiding frequency.
Level of agreement nighttime voided volume versus nighttime voiding frequency | Through study completion, an average of 1.5 year
  What are the mean differences and the limits of agreement between the pBD and autoBD for nighttime voided volume versus nighttime voiding frequency.
Patient compliance reported by patient | Through study completion, an average of 1.5 year
  Subjective compliance will be assessed using topics such as completion, reliability, time to data entry, measuring accuracy, child involvement, child's and parents' motivation and interference with daily life.
Patient compliance reported by healthcare provided | Through study completion, an average of 1.5 year
  Subjective compliance will be assessed using topics such as completion, measuring accuracy, quality, reliability and clinical usefulness
Patient satisfaction | Through study completion, an average of 1.5 year
  Patient satisfaction will be assessed on usability, ergonomics, and diary preference.
Healthcare professional satisfaction | Through study completion, an average of 1.5 year
  Healthcare professional satisfaction will be assessed on user experience related to setting up and interpreting the diaries and diary preference.
  Healthcare professional satisfaction will be assessed on user experience related to setting up and interpreting the diaries and diary preference.

CONTACTS AND LOCATIONS:
Overall Officials: Gunter De Win, PhD, Principal Investigator — UZA/UAntwerpen
Locations (5):
- Belgium (5):
  - UZA, Edegem, Antwerpen
  - AZ Voorkempen, Malle, Antwerpen
  - Imelda Ziekenhuis, Bonheiden, Antwerp
  - Privé praktijk dr. Katrien Klockaerts, Aalst, Oost-Vlaanderen
  - ZNA Koningin Paola Kinderziekenhuis, Antwerp

IPD SHARING:
Plan to Share IPD: No